CLINICAL TRIAL: NCT01008943
Title: A Canadian Prospective Nonrandomized Study of Autologous Cell Therapy for Female Stress Urinary Incontinence
Brief Title: Autologous Cell Therapy for Female Stress Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-013
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Autologous Muscle Derived Cells

INTERVENTIONS:
Biological: Autologous Muscle Derived Cells — Urethral injection of autologous muscle-derived cells

SUMMARY:
The Autologous Cell Therapy for Female SUI study is a clinical trial to determine the safety and potential effectiveness of a single dose of 200 million Cook MyoSite Autologous Muscle Derived Cells for treatment of Stress Urinary Incontinence.

ELIGIBILITY:
Inclusion Criteria:

* SUI with normal detrusor activity confirmed with urodynamics
* Bladder capacity >200 ml
* Incontinence has not shown any improvement for at least -6 months
* Failed prior treatments (e.g., behavior modification, bladder exercises, biofeedback, electrical stimulation, bulking injections, urethral suspensions and/or drug therapy)

Exclusion Criteria:

* Known vesicoureteral reflux, vaginal prolapse beyond the introitus, or other significant pelvic floor abnormalities with high pressure instability
* Neuromuscular disorder (e.g., muscular dystrophy, multiple sclerosis)
* Uncontrolled diabetes
* Pregnant, lactating, or plans to become pregnant during course of the study
* Morbid obesity (defined as 100 pounds over their ideal body weight, or BMI ≥40) and not expected to benefit from treatment
* Current or acute conditions involving cystitis or urethritis
* Scheduled to receive radiation treatment to the vicinity, or history of radiation treatment to the urethra or adjacent structures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06-02 (Actual); Primary Completion 2012-09-21 (Actual); Study Completion 2012-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley K. Carr, MD, Principal Investigator — Sunnybrook Health Sciences Center
Locations (2):
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - Sunnybrook Health Sciences Center, Toronto, Ontario

REFERENCES:
- See also: Autologous muscle derived cells for treatment of stress urinary incontinence in women — http://www.ncbi.nlm.nih.gov/pubmed/24582537

RESULTS

PARTICIPANT FLOW:
Groups:
- Autologous Muscle-Derived Cells (AMDC): Intrasphincteric injection of 200 million AMDC for treatment of SUI in women
Period: Overall Study
Arm/Group | Autologous Muscle-Derived Cells (AMDC)
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Autologous Muscle-Derived Cells (AMDC)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced Biopsy Procedure-related Adverse Events
Description: Biopsy was required to generate AMDC products. Biopsy procedure-related events were defined as systemic responses to the biopsy procedure or injury at the biopsy site. Since biopsy occurred prior to AMDC treatment, results are presented independent of AMDC dose received. All biopsy procedure-related events either self-resolved or were easily treated.
Time Frame: at biopsy or between biopsy and treatment, approximately 6 weeks
Population: One patient experienced procedural dizziness.
Measure: Number; unit: participants
Units Other Than Participants: Biopsies
Arm/Group | Autologous Muscle-Derived Cells (AMDC)
Number analyzed (Participants) | 16
Number analyzed (Biopsies) | 22
participants | 1

2. Primary Outcome: Number of Participants That Experienced Injection Procedure-related Adverse Events
Description: AMDC treatment was administered via intrasphincteric injection. Injection procedure-related events were defined as systemic responses to the injection procedure or genitourinary events occurring within 30 days of the injection procedure that could be attributed to cystoscopy or catheterization. Since these events could be attributed to the injection procedure, results are considered independent of AMDC dose received. All injection procedure-related events self-resolved or were easily treated.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Autologous Muscle-Derived Cells (AMDC)
Number analyzed (Participants) | 16
participants | 6

3. Primary Outcome: Injection Procedure-related Adverse Events
Description: as for outcome 2
Time Frame: 30 days
Measure: Number; unit: events
Arm/Group | Autologous Muscle-Derived Cells (AMDC)
Number analyzed (Participants) | 16
events
  Abdominal pain lower | 2
  Dysuria | 4
  Micturition urgency | 1
  Urinary tract infection | 1

4. Primary Outcome: Number of Participants That Experienced AMDC Product-related Events
Description: If an immune response after injection or any urinary retention occurred and seemed suspicious, the physicians were consulted to determine whether the effect was likely related to the AMDC product.
  No adverse events reported during the study were adjudicated as AMDC product-related.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Autologous Muscle-Derived Cells (AMDC)
Number analyzed (Participants) | 16
participants | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Autologous Muscle-Derived Cells (AMDC)
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Muscle-Derived Cells (AMDC) (N=16)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) — Patient fractured the proximal end of fibula when fell horse-riding, which required medical intervention and resulted in persistent or significant disability or incapacity. It was adjudicated as not related to study procedures or AMDC treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Muscle-Derived Cells (AMDC) (N=16)
After AMDC treatment: Abdominal pain lower (Gastrointestinal disorders) | 2 (2)
After AMDC treatment: Generalised oedema (General disorders) | 1 (1)
After biopsy, before AMDC: Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1)
After AMDC treatment: Blood creatinine increased (Investigations) | 1 (1)
After AMDC treatment: Blood urea increased (Investigations) | 1 (1)
After AMDC treatment: Blood urine (Investigations) | 1 (1)
After AMDC treatment: Hemoglobin decreased (Investigations) | 1 (1)
After AMDC treatment: Platelet count decreased (Investigations) | 1 (1)
After AMDC treatment: Protein urine present (Investigations) | 1 (1)
After AMDC treatment: Residual urine volume increased (Investigations) | 1 (1)
After AMDC treatment: White blood cell count increase (Investigations) | 2 (2)
After AMDC treatment: Dysuria (Renal and urinary disorders) | 5 (5)
After AMDC treatment: Micturition urgency (Renal and urinary disorders) | 1 (1)
After biopsy, before AMDC: Urethral dilatation (Renal and urinary disorders) | 1 (1) — Urethra dilated immediately proceding the injection procedure to allow passage of the needle into the urethra.
After AMDC treatment: Urinary retention (Renal and urinary disorders) | 2 (2)
After AMDC treatment: Urinary tract infection (Renal and urinary disorders) | 3 (3)
After AMDC treatment: Menorrhagia (Reproductive system and breast disorders) | 1 (1)
After AMDC treatment: Menstruation irregular (Reproductive system and breast disorders) | 1 (1)
After AMDC treatment: Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1)
After AMDC treatment: Ophthalmologic treatment (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days